CLINICAL TRIAL: NCT06202183
Title: Exercise for Gut Microbiome in Patients With Young-Onset Colorectal Cancer Undergoing Chemotherapy: The COURAGE Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-341
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; Metastatic Colon Cancer; Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Metastatic Colon Cancer; Metastatic Colorectal Cancer; Early Stage Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Masking Description: blinded to block size
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Exercise Group (Experimental): 42 participants will be enrolled using a permuted blocked design with varying block size and will complete study procedures as follows:
  * Baseline in-office visit.
  * Completion of exercise sessions 3x weekly.
  * Post-intervention in-office visit.
  Interventions: Behavioral: Exercise Program
- Group B: Waitlist Control Group (No Intervention): 42 participants will be enrolled using a permuted blocked design with varying block size and will complete study procedures as follows:
  * Baseline in-office visit.
  * Participants will be asked to maintain baseline exercise behavior and/or usual, daily activities.
  * Post-intervention in-office visit. Participants will be offered to participate in the exercise program upon the completion of post-intervention assessments.

INTERVENTIONS:
Behavioral: Exercise Program — A 12 week, home-based, virtually supervised, aerobic and resistance exercise training program comprised of 36 sessions. Participants will be provided with a home stationary bike, resistance bands, and Fitbit. Virtually supervised sessions will be accessible via Zoom platform. For participants who do not have a device, a Wi-Fi-enabled tablet will also be provided.
  Arms: Group A: Exercise Group

SUMMARY:
This research study is a randomized controlled trial that will observe changes in microbiome activity, changes in chemotherapy toxicity, and any changes in treatment outcomes between two groups of participants undergoing chemotherapy with either early-stage or metastatic colorectal cancer.

The names of the study groups involved in this study are:

* Exercise
* Waitlist Control

DETAILED DESCRIPTION:
This research study is a single-center, two-armed, randomized controlled trial that will observe changes in microbiome activity, changes in chemotherapy toxicity, and any changes in treatment outcomes between two groups of participants undergoing chemotherapy with either early-stage or metastatic colorectal cancer. Participants will be randomly assigned to one of two groups: Group A: Exercise group (EXE) vs. Group B: Waitlist control group (WC). Randomization means that a participant will be placed into one of the study groups by chance.

The research study procedures include screening for eligibility, blood tests, stool samples, and survey questionnaires.

Participation in this research study will last up to 6 months.

It is expected that about 84 people will take part in this research study.

The American Cancer Society is providing funding for this research study.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with early-stage or metastatic colon or rectal cancer
* Age at diagnosis 18-50 years; due to the specificity of the study question those outside the age bracket will not be included
* No plans for major surgical intervention at the time of recruitment for a minimum of 12 weeks (i.e. study period; placement of port a cath is allowed)
* No plans for radiation therapy at the time of recruitment for a minimum of 12 weeks
* On or planning chemotherapy
* Participate in less than or equal to 90 minutes of moderate-to-vigorous exercise per week
* Medical clearance to perform exercise intervention and testing by their treating oncologist
* No uncontrolled medical conditions that could be exacerbated with exercise
* Ability to communicate and complete written forms in English
* Ability to understand and the willingness to sign informed consent prior to any study-related procedures
* Willing to travel to DFCI for necessary data collection

Exclusion Criteria:

* Participate in more than 90 minutes of moderate-to-vigorous aerobic exercise per week over the past month. This study targets insufficiently active persons to assess the effect of the described exercise intervention, where additional exercise done regularly will contaminate the intervention effects.
* Unstable comorbidities that prevent participation in moderate-to-vigorous intensity exercise. Patients with unstable comorbidities may develop unexpected adverse events from exercise. For the purpose of patients' safety, as well as because this study involves remote, home-based exercise where close supervision is not possible, patients with unstable medical conditions are excluded.
* Patients actively on a weigh loss diet and/or actively taking weight loss drugs. This could effect gut microbiome.
* Patient with other active malignancies (excluding basal cell carcinoma).
* Subjects who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome Genomes | Baseline (Week 1) and Post-intervention (Week 13)
  Gut Microbiome Sequencing will be conducted using the stool samples at Baseline and Post-Intervention. Gut Microbiome sequencing will be performed using DNA and RNA extraction, which will analyze microbial genomes.

SECONDARY OUTCOMES:
Change in Chemotherapy Toxicity | 12 weeks
  To evaluate changes in chemotherapy toxicity following a exercise intervention in survivors of young-onset CRC undergoing chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, MPH, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu